CLINICAL TRIAL: NCT02835638
Title: Observational Multicenter Cohort Study of French Patients With a Central or Combined Syndrome of Sleep Apnea With a Predominant Central SAS Treated by Adaptive Servo-Ventilation
Brief Title: Quality of Sleep of Patients With Predominant Central Sleep Apnea Syndrome(SAS) Whose EF > 45% Treated by ASV
Acronym: FACIL-VAA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Société Française de Recherche et de Médecine du Sommeil (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-A01186-45
Record Dates: First submitted 2016-07-08; First posted 2016-07-18 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2022-09

CONDITIONS: Central Sleep Apnea Syndrome in Patients Whose EF is Above 45 Percent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Adaptative Servo Ventilation — the ASV treatment will be observed during this study on the patients included

SUMMARY:
The main goal of this French multicenter observational cohort study is to prospectively collect data assessing the impact of the Adaptative Servo-Ventilation treatment on the quality of sleep of patients with central or combined sleep apnea syndrome (SAS) out of Heart Failure (HF) with altered ejection fraction, with a predominant central SAS.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years
* Naive patient to treatment with positive pressure with AHIc > 15 requiring the establishment of an ASV to a central or combined SAS without any systolic HF (LVEF ≤ 45%) with predominant central SAS.

  * OR Patient with a predominant obstructive SAS ( ≤ 50% central event ) whose Continuous Positive Airway Pressure treatment (CPAP) does not allow adequate control of the central events: treated for at least 1 month CPAP with a residual central apnea hypopnea index greater than or equal to 10 events per hour (AHI global> 15, which AHIc ≥ 10) pressure to control obstructive events ( IAHo <5 ) controlled by polygraphy or polysomnography with a pressure test <10 cm H2O.
* Before inclusion, for patients who have previously been treated with CPAP, a PSG diagnosis will be made after a period of wash-out of CPAP of a 1-week period.
* Patient affiliated to the national social security (beneficiary or assignee ).
* Patient being aware of the information form and signed informed consent.

Exclusion Criteria:

* Patients with against -indication for the use of ASV :

  * History of massive epistaxis.
  * Diseases related to barotrauma particularly pneumothorax and pneumo- mediastinum.
  * Suspicions of meningeal gaps or trauma history of the prior stage of the skull base.
  * Shortness of breath or hypercapnia deemed incompatible by the doctor with the ASV treatment.
* Patients with predominant obstructive sleep apnea (OSA) (> 85% obstructive events ).
* Standardized central SAS by the Continuous Positive Airway Pressure
* Patients with a diagnosis of systolic heart failure (LVEF ≤45 %) with a predominant central SAS ( > 50% central events ).
* Person deprived of liberty by judicial or administrative decision, person under a legal protection measure (pregnant or lactating women, patients under guardianship)
* Lack of signature for the information form and the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Central or Combined Sleep Apnea Syndrome (SAS) Out of Heart Failure (HF) With Altered Ejection Fraction, With a Predominant Central SAS.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
quality of sleep | 6 months
  assessment of the evolution of the sleep quality using the Pittsburgh Sleep Quality Index ( PSQI ) in all patients for any etiologies.

CONTACTS AND LOCATIONS:
Locations (28):
- France (28):
  - CHU de Poitiers, Poitiers, Nouvelle-Aquitaine
  - CHU d'Angers, Angers
  - CH Antibes, Antibes
  - Centre Hospitalier de Béziers, Béziers
  - Hôpital de Chantilly Les Jockeys, Chantilly
  - Hôpital Antoine Béclère, Clamart
  - Hôpital Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - Groupe Hospitalier La Rochelle Ré Aunis, La Rochelle
  - CH du Mans, Le Mans
  - Clinique La Louvière, Lille
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Hôpital Arnaud de Villeneuve CHU de Montpellier, Montpellier
  - Groupe Hospitalier de la Région de Mulhouse et Sud Alsace, Mulhouse
  - Hôpital Universitaire Saint Antoine, Paris
  - Hôpital Bichat, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - CH Annecy Annecy, Pringy
  - Hôpital Maison Blanche CHU de Reims, Reims
  - Cabinet Libéral de Pneumologie, Rennes
  - Centre VISAS, Saint-Etienne
  - Groupe Hospitalier Public du Sud de l'Oise, Senlis
  - Cabinet Libéral Selest, Strasbourg
  - CHU de Strasbourg, Strasbourg
  - Hôpital Larrey, Toulouse
  - CHU de Nancy, Vandœuvre-lès-Nancy
  - Centre Hospitalier Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: Yes
oversight committee

REFERENCES:
- [Derived] Tamisier R, Philippe C, Prigent A, Charley-Monaca C, d'Ortho MP, Gentina T, Gagnadoux F, Launois C, Bironneau V, Mallet JP, Didi T, Guy T, Goutorbe F, Perrin C, Pontier-Marchandise S, Timsit JF, Pepin JL, Meurice JC; Etude de Cohorte Observationnelle Multicentrique Francaise de Patients Ayant un Syndrome d'Apnees du Sommeil Central ou Combine Avec SAS Central Predominant, Traites par Ventilation Auto-asservie Investigators. Change in Sleep Quality Associated With Adaptive Servoventilation for Central Sleep Apnea: Six-Month Follow-Up of the Multicenter Nationwide French "Etude de Cohorte Observationnelle Multicentrique Francaise de Patients Ayant un Syndrome d'Apnees du Sommeil Central ou Combine Avec SAS Central Predominant, Traites par Ventilation Auto-Asservie (FACIL-VAA)" Cohort. Chest. 2025 Apr;167(4):1204-1217. doi: 10.1016/j.chest.2024.12.015. Epub 2024 Dec 20. PMID 39710250
- See also: Description of the previous study SERVE-HF that included only altered LVEF patients. The SERVE-HF's population is the one the FACIL-VAA study is avoiding. — http://www.resmed.com/us/en/consumer/newsandinformation/news-releases/2015/resmed-provides-update-on-phase-iv-serve-hf-study-of-adaptive-servo-ventilation-therapy.html